CLINICAL TRIAL: NCT01427634
Title: Randomized Controlled Trial of Proactive Palliative Care for Patients With Ventricular Assist Devices and Their Families
Brief Title: Proactive Palliative Care for Patients With Ventricular Assist Devices (VAD) and Their Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH); The Greenwall Foundation (Unknown); Emily Davie and Joseph S. Kornfeld Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GCO 11-0152; P30AG028741-01A2 (NIH)
Record Dates: First submitted 2011-08-15; First posted 2011-09-01 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Heart Failure; End-stage Disease
Keywords: Heart Failure; Ventricular Assist Device; Palliative Care
MeSH Terms: conditions — Heart Failure | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palliative Care (Active Comparator): Receive ongoing counseling and symptom assessment as well as clarification and documentation of goals of care, starting before implantation and continuing throughout the course of the study. Intervention patients will also be followed by the inpatient palliative care consultation service when hospitalized for their initial VAD implantation and during any subsequent hospitalizations as needed
  Interventions: Behavioral: Palliative Care
- Control (Other): Usual Care
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Palliative Care — Receive ongoing counseling and symptom assessment as well as clarification and documentation of goals of care, starting before implantation and continuing throughout the course of the study. Intervention patients will also be followed by the inpatient palliative care consultation service when hospitalized for their initial VAD implantation and during any subsequent hospitalizations as needed
  Arms: Palliative Care
Other: Usual Care — Receive usual care as provided by the VAD clinical team.
  Arms: Control

SUMMARY:
The primary aim of the study is to provide "proof of concept" to demonstrate that patients with Ventricular Assist Devices (VADs) and caregivers are willing to be enrolled in a randomized trial of palliative care and that such a study is feasible. Secondary aims include demonstrating improvement in symptoms (physical and psychological) for intervention patients and their caregivers as compared to control patients and caregivers. The investigators will also examine differences in utilization of healthcare services, mortality, and completion of advance directives between intervention and control patients.

DETAILED DESCRIPTION:
A ventricular assist device is an implanted mechanical device which augments the pumping function of the heart's ventricles. The number of patients with VADs is expected to increase in an exponential manner in the years to come as device technology improves and continues to show a survival benefit. The investigators propose a randomized controlled trial of a proactive palliative care intervention for patients with VADs and their caregivers. Patients randomized to palliative care will receive ongoing counseling and symptom assessment as well as clarification and documentation of goals of care, starting before implantation and continuing throughout the course of the study. The intervention is delivered primarily in the outpatient setting by a palliative care nurse practitioner. Intervention patients will also be followed by the inpatient palliative care consultation service when hospitalized for their initial VAD implantation and during any subsequent hospitalizations as needed. Control patients will receive usual care as provided by the VAD clinical team. Data collection will be performed by a research assistant at Mount Sinai (blinded to randomization) who conducts baseline assessments in person, and then follow-up assessments over the phone. The primary aim of the study is to provide "proof of concept" to demonstrate that patients and caregivers are willing to be enrolled in a randomized trial of palliative care and that such a study is feasible. Secondary aims include demonstrating improvement in symptoms (physical and psychological) for intervention patients and their caregivers as compared to control patients and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* age >21 years
* fluent in English
* have a caregiver/family member who is willing to be enrolled and who is also fluent in English
* consistent and reliable access to a phone

Exclusion Criteria:

* non English-speaking

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Pain Assessment - change at 1 year from baseline | baseline (within 2 weeks of enrollment) and at 1 year after implantment
  change in pain from baseline to 1 year, using the Memorial Symptom Assessment Scale

SECONDARY OUTCOMES:
Satisfaction with care - change at 1 year from baseline | at baseline (within 2 weeks of enrollment) and at 1 year after implantment
  changes in satisfaction with care from baseline to 1 year as measured with validated scales for satisfaction with care.
PROMIS anxiety scale - change at 1 year from baseline | at baseline (within 2 weeks of enrollment) and at 1 year after implantment
  changes in anxiety from baseline to 1 year as measured by the PROMIS anxiety scale
PROMIS depression scale - change at 1 year from baseline | at baseline (within 2 weeks of enrollment) and at 1 year after implantment
  changes in depression measured from baseline to 1 year as measured by the PROMIS depression scale

CONTACTS AND LOCATIONS:
Overall Officials: Nathan E. Goldstein, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] WRITING GROUP MEMBERS; Lloyd-Jones D, Adams RJ, Brown TM, Carnethon M, Dai S, De Simone G, Ferguson TB, Ford E, Furie K, Gillespie C, Go A, Greenlund K, Haase N, Hailpern S, Ho PM, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott MM, Meigs J, Mozaffarian D, Mussolino M, Nichol G, Roger VL, Rosamond W, Sacco R, Sorlie P, Roger VL, Thom T, Wasserthiel-Smoller S, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2010 update: a report from the American Heart Association. Circulation. 2010 Feb 23;121(7):e46-e215. doi: 10.1161/CIRCULATIONAHA.109.192667. Epub 2009 Dec 17. No abstract available. PMID 20019324
- [Background] Kirklin JK, Naftel DC, Kormos RL, Stevenson LW, Pagani FD, Miller MA, Ulisney KL, Baldwin JT, Young JB. Second INTERMACS annual report: more than 1,000 primary left ventricular assist device implants. J Heart Lung Transplant. 2010 Jan;29(1):1-10. doi: 10.1016/j.healun.2009.10.009. No abstract available. PMID 20123242